CLINICAL TRIAL: NCT00338611
Title: Convergence Insufficiency Treatment Trial (CITT)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Mitchell Scheiman, OD, Pennsylvania College of Optometry
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEI-107
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2008-10

CONDITIONS: Convergence Insufficiency; Binocular Vision Disorder
Keywords: vision therapy; orthoptics; pencil push-up therapy
MeSH Terms: conditions — Ocular Motility Disorders | interventions — Orthoptics

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Behavioral: Home-based Pencil Push-Up Therapy — Exercise in which patients visually followed a small letter on a pencil as they moved the pencil closer to the bridge of their nose
Behavioral: Home-based Pencil Push-ups with Computer Vision Therapy/Orthoptics — Exercise in which patients visually followed a small letter on a pencil as they moved the pencil closer to the bridge of their nose combined with additional computer vision therapy
Behavioral: Office-based Vision Therapy/Orthoptics — Weekly hour-long sessions of office-based vision therapy with a trained therapist and performed at-home reinforcement exercises
Behavioral: Placebo Office-based Vision Therapy/Orthoptics — Vision activities designed to simulate office-based therapy

SUMMARY:
The purposes of the CITT are:

* To determine whether Home-based Pencil Push-up therapy, Home-based Pencil Push-ups with Computer Vision Therapy/Orthoptics or Office-based VT/Orthoptics more effective than placebo treatment, and whether there are differences between the three treatments in improving subject symptoms and signs.
* To evaluate whether improvements in outcome measures are still present after one year of observation.

DETAILED DESCRIPTION:
Convergence insufficiency is a prevalent and distinct binocular vision disorder. Typical symptoms include double vision, eyestrain, headaches, and blurred vision while reading. It affects approximately 5% of children in the United States, and may have a serious impact on an individual's performance in school, choice of jobs, and quality of life.

There is no consensus regarding the most effective treatment for convergence insufficiency. Two commonly prescribed treatments are home-based pencil push-up therapy and office-based vision therapy/orthoptics. Significant differences exist between these two treatment modalities in cost and number of office visits required, with pencil push-up therapy being less expensive and less time intensive. There have been no well-designed studies that have compared the effectiveness of these two treatments.

The Convergence Insufficiency Treatment Trial (CITT) is a prospective, masked, placebo-controlled, multi-center clinical trial in which 208 subjects between the ages of 9 to < 18 years will be randomly assigned to: 1) Home-based Pencil Push-Up Therapy, 2) Home-based Pencil Push-ups with Computer Vision Therapy/Orthoptics, 3) Office-based Vision Therapy/Orthoptics, or 4) Placebo Office-based Vision Therapy/Orthoptics. The primary outcome measure is a measure of symptoms using a 15-item survey, the CI Symptom Survey. Secondary outcome measures are two common clinical tests of the eyes' ability to converge when performing close work. Patients will be tested at the eligibility examination, and by masked examiners after 4, 8 and 12 weeks of treatment have been completed during the 12-week treatment phase. Long term follow-up will be assessed at 6 and 12 months after the completion of active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 9 and 17 years with symptomatic convergence insufficiency
* Exophoria at near at least 4Δ greater than at far
* Insufficient positive fusional convergence at near
* A receded near point of convergence of ≥6 cm break
* CI Symptom Survey score ≥16

Exclusion Criteria:

* Previous treatment with office-based vision therapy/orthoptics or pencil push-ups
* Systemic diseases known to affect accommodation, vergence and ocular motility
* Developmental disability, mental retardation, attention deficit hyperactivity disorder (ADHD), or learning disability diagnosis that in the investigator's discretion would interfere with treatment

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 221 (Actual)
Dates: Start 2005-07; Primary Completion 2008-09 (Actual); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Measure of symptoms using a 15-item Convergence Insufficiency Symptom Survey | 12 weeks

SECONDARY OUTCOMES:
Eyes' ability to converge when performing close work | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Scheiman, OD, Study Chair — Pennsylvania College of Optometry
Locations (9):
- United States (9):
  - University of Alabama at Birmingham School of Optometry, Birmingham, Alabama
  - Southern California College of Optometry, Fullerton, California
  - Ratner Children's Eye Center, La Jolla, California
  - NOVA Southeastern University College of Optometry, Fort Lauderdale, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Mayo Clinic, Rochester, Minnesota
  - State University of New York College of Optometry, New York, New York
  - The Ohio State University College of Optometry, Columbus, Ohio
  - Pennsylvania College of Optometry, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Convergence Insufficiency Treatment Trial Study Group. Randomized clinical trial of treatments for symptomatic convergence insufficiency in children. Arch Ophthalmol. 2008 Oct;126(10):1336-49. doi: 10.1001/archopht.126.10.1336. PMID 18852411
- [Derived] Scheiman M, Kulp MT, Cotter SA, Lawrenson JG, Wang L, Li T. Interventions for convergence insufficiency: a network meta-analysis. Cochrane Database Syst Rev. 2020 Dec 2;12(12):CD006768. doi: 10.1002/14651858.CD006768.pub3. PMID 33263359
- [Derived] CITT-ART Investigator Group. Treatment of Symptomatic Convergence Insufficiency in Children Enrolled in the Convergence Insufficiency Treatment Trial-Attention & Reading Trial: A Randomized Clinical Trial. Optom Vis Sci. 2019 Nov;96(11):825-835. doi: 10.1097/OPX.0000000000001443. PMID 31651593
- [Derived] Barnhardt C, Cotter SA, Mitchell GL, Scheiman M, Kulp MT; CITT Study Group. Symptoms in children with convergence insufficiency: before and after treatment. Optom Vis Sci. 2012 Oct;89(10):1512-20. doi: 10.1097/OPX.0b013e318269c8f9. PMID 22922781
- [Derived] Scheiman M, Kulp MT, Cotter S, Mitchell GL, Gallaway M, Boas M, Coulter R, Hopkins K, Tamkins S; Convergence Insufficiency Treatment Trial Study Group. Vision therapy/orthoptics for symptomatic convergence insufficiency in children: treatment kinetics. Optom Vis Sci. 2010 Aug;87(8):593-603. doi: 10.1097/OPX.0b013e3181e61bad. PMID 20543758
- [Derived] Rouse M, Borsting E, Mitchell GL, Kulp MT, Scheiman M, Amster D, Coulter R, Fecho G, Gallaway M; CITT Study Group. Academic behaviors in children with convergence insufficiency with and without parent-reported ADHD. Optom Vis Sci. 2009 Oct;86(10):1169-77. doi: 10.1097/OPX.0b013e3181baad13. PMID 19741558
- [Derived] Convergence Insufficiency Treatment Trial Study Group. Long-term effectiveness of treatments for symptomatic convergence insufficiency in children. Optom Vis Sci. 2009 Sep;86(9):1096-103. doi: 10.1097/OPX.0b013e3181b6210f. PMID 19668097
- [Derived] Kulp M, Mitchell GL, Borsting E, Scheiman M, Cotter S, Rouse M, Tamkins S, Mohney BG, Toole A, Reuter K; Convergence Insufficiency Treatment Trial Study Group. Effectiveness of placebo therapy for maintaining masking in a clinical trial of vergence/accommodative therapy. Invest Ophthalmol Vis Sci. 2009 Jun;50(6):2560-6. doi: 10.1167/iovs.08-2693. Epub 2009 Jan 17. PMID 19151384